CLINICAL TRIAL: NCT04907981
Title: Risk Screening Based on Feature Recognition and Detection of Eye Surface Images of COVID-2019 Patients and Statistical Analysis of High-dimensional Data
Brief Title: Eye Detection to Identify Novel Coronavirus Infection
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Fudan University (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Fifth Hospital of Shijiazhuang City (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19
Record Dates: First submitted 2021-05-23; First posted 2021-06-01 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Novel coronavirus infection: All patients were diagnosed according to the diagnostic criteria of the National Health Commission of China and confirmed by RT-PCR detection of viral nucleic acids.
  Interventions: Diagnostic Test: Novel coronavirus infection
- Not infected by novel coronavirus: Healthy controls and patients with liver disease
- Recovered patients with nucleic acid negative after infection with novel coronavirus: Novel coronavirus nucleic acid changed from positive to negative.

INTERVENTIONS:
Diagnostic Test: Novel coronavirus infection — Using eye examination to judge whether novel coronavirus is infected or not.
  Groups: Novel coronavirus infection

SUMMARY:
The eye characteristics of patients with COVID-19 and those without the disease were analyzed, and whether they had the disease or not was judged according to the eye characteristics.

DETAILED DESCRIPTION:
To test the accuracy of a non-invasive eye monitoring that can be widely used for screening in judging patients with novel coronavirus infection.

ELIGIBILITY:
Inclusion Criteria:

1. All participants were provided with written informed consent at the time of recruitment；
2. Age ≥ 18 and ≤ 75 (informed consent signed by guardian under 18)
3. Meet the diagnostic criteria of novel coronavirus (2019-COVID-19) infection

Exclusion Criteria:

Does not meet any of the inclusion criteria

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Collection and analysis of eye characteristics of patients encoding criteria, annotation of ocular feature | 1DAY
  Ocular pathological features

CONTACTS AND LOCATIONS:
Overall Officials: Lei zhao, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Shijiazhuang Fifth Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided